CLINICAL TRIAL: NCT02566434
Title: Methionine Tolerance in Healthy Human Adults
Acronym: Met
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: International Council on Amino Acid Science (Other)
Responsible Party: Principal Investigator, Marielle PKJ Engelen, PhD, Associate Professor, Texas A&M University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-0800
Record Dates: First submitted 2015-09-21; First posted 2015-10-02 (Estimated); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: Dietary Supplements
MeSH Terms: interventions — Methionine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methionine (Experimental): All participants will consume free methionine at 10 mg/kg body weight/day (=requirement), 25 mg/kg body weight/day, 50 mg/kg body weight/day and 100 mg/kg body weight/day for the duration of a 4-week intervention period. Participants will cease intake when signs of toxicity are measured in blood work.
  Interventions: Dietary Supplement: methionine

INTERVENTIONS:
Dietary Supplement: methionine — 4 weeks intervention and 2 to 4 weeks washout in healthy volunteers with free methionine at 10 mg/kg body weight/day (=requirement), 25 mg/kg body weight/day, 50 mg/kg body weight/day and 100 mg/kg body weight/day.

SUMMARY:
Participants will receive four different doses of methionine through four month long interventions with a two week wash-out period in between intervention. The dose will increase with each intervention. Two visits during each intervention will also involve receiving stable isotope infusion to determine the metabolism of methionine in the body. Participants will also be monitored via blood work and questionnaires regarding overall health.

DETAILED DESCRIPTION:
Study subjects: Healthy volunteers (40 - 79 years) will be included in the study. Informed consent will be obtained before any study related procedures will be performed. All subjects will be extensively screened by research nurses / physician. Exclusion criteria are any condition that interfere with the definition 'healthy" according to the study physician's judgement based on medical history, lab testing, use of medication, and physical exam.

Study design: To establish the Upper Level of Safe intake (USLI) of methionine intake, it is essential to create a dose-response approach of possible negative effects of methionine. To define the Lowest-Observed-Adverse-Effect Level (LOAEL), the investigators suggest a 4 weeks intervention and 2 to 4 weeks washout in healthy volunteers with free methionine at 10 mg/kg body weight/day (=requirement), 25 mg/kg body weight/day, 50 mg/kg body weight/day and 100 mg/kg body weight/day. Pure methionine will be provided by ICAAS. The 4-week intervention period is based on a study in pigs (6). Methionine will be consumed in 3 daily doses. Participants will be advised about their daily dietary intake during the study. Besides the screening visit, each subjects will come back for up to 13 study visits (up to 5 Short study Days (SD, approx. 30 min) and 8 Long study Days (LD, approx. 5 h). On all study days (both SD and LD) the investigators will check parameters of toxicity and measure metabolites of methionine catabolism on the day before each dose intervention, during intervention (2 weeks after the start of each dose intervention; range: +/- 3 days), on the last day of each dose intervention, and 2 weeks after the last dose intervention. Because methionine as a dietary supplement clearly rises a safety issue, we will conduct this experiment in steps. First, subjects will receive the 10 mg/kg body weight/day. The investigators then will analyse all parameters of toxicity, interpret the data and when there are no safety concerns, continue with the next intake level. The study will be stopped at the level when there are apparent safety concerns.

The study will take place at the research facility of the Center for Translational Research on Aging and Longevity (CTRAL), Texas A&M University. The subject will be asked to arrive in the fasted state on both the screening and all study days. On the screening day, body weight and height will be measured and Dual-energy X-ray absorptiometry (DXA) will be performed to measure body composition. On both SD and LD a medical interview will be performed and a toxicity questionnaire completed (see attached protocol). Furthermore on a SD two blood samples will be taken (up to 30 ml). On a LD, one catheter will be inserted in the peripheral vein of an arm for blood sampling (18 samples in total, up to 80 ml per LD) and questionnaires related to cognition, health status and well being may or may not be completed by the subject (see attached protocol). After a baseline blood sample is taken, a stable isotope pulse is provided through the same line. The baseline sample will be used to test toxicity parameters in blood, plasma homocysteine concentration, the plasma concentrations of products of the methionine degrading transamination and sulfoxidation route, and to establish background enrichment of stable isotopes. Samples obtained after the pulse will provide information about transmethylation of methionine, and GSH synthesis. Subjects will be called every week to check compliance regarding supplement intake and to answer questions regarding health and well-being. Subjects who discontinue the study during the study will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a healthy male or female according to the investigator's or appointed staff's judgment
2. Age 40 - 79 years.
3. Must be willing to lay in bed for 4 hours on the long study days (LD)
4. Have a stable body weight within the past 3 months (< 5% change)

Exclusion Criteria:

1. History of cardiovascular disease
2. Metabolic diseases including hepatic or renal disorder
3. Presence of acute illness or metabolically unstable chronic illness
4. Unwilling to stop taking nutritional supplements containing proteins or free amino acids within 5 days of the first study day until study completion
5. Have not taken or participated in any nutritional supplement study program within the past 4 weeks
6. Any other condition according to the PI or nurse that would interfere with the study or safety of the subject or influence the results
7. Pregnancy
8. Unwilling to comply with any other rules set forth in the Informed Consent Form

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2016-04 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Hepatic Function Panel--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Metabolic Renal Function Panel--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Blood Count (CBC) With Differential--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Hepatic Function Panel--25 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Metabolic Renal Function Panel--25mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Blood Count (CBC) With Differential--25 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Hepatic Function Panel--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Metabolic Renal Function Panel--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Blood Count (CBC) With Differential--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Hepatic Function Panel--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Metabolic Renal Function Panel--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Blood Count (CBC) With Differential--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks

SECONDARY OUTCOMES:
Complete Aminogram--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Glutathione ratio--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Plasma Homocysteine concentration--10 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Aminogram--25 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Glutathione ratio--25 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Plasma Homocysteine concentration--25 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Aminogram--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Glutathione ratio--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Plasma Homocysteine concentration--50 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Complete Aminogram--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Glutathione ratio--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks
Plasma Homocysteine concentration--100 mg/kg body weight dose | participants will be followed for the duration of the dose intervention, an expected average of 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Engelen, Study Director — Texas A&M University
Locations (1):
- Texas A&M University-CTRAL, College Station, Texas, United States

REFERENCES:
- [Derived] Deutz NE, Simbo SY, Ligthart-Melis GC, Cynober L, Smriga M, Engelen MP. Tolerance to increased supplemented dietary intakes of methionine in healthy older adults. Am J Clin Nutr. 2017 Aug;106(2):675-683. doi: 10.3945/ajcn.117.152520. Epub 2017 Jun 21. PMID 28637772